CLINICAL TRIAL: NCT06176014
Title: Effect of Using Polyetherketoneketone (PEKK) Framework Versus Cobalt Chromium Framework on The Supporting Structures of Mandibular Implant Supported Hybrid Prostheses
Brief Title: Effect of Using (PEKK) Framework Versus (Co- Cr) Framework on The Bone of Mandibular Implant Supported Hybrid Prostheses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FDASU-RecID032134
Record Dates: First submitted 2023-12-07; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Alveolar Bone Loss
Keywords: hybrid prosthesis; PEKK framework; PFM framework
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: to compare PEKK framework for hybrid prostheses ( fixed detachable ) versus PFM framework
Who Masked: Investigator
Masking Description: all the selected patients were rehabilitated with lower single denture then divided by computer randomization using random allocation software
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (PEKK fixed hybrid prostheses (Other): 5 implants were placed in mandibular arch by surgical guide and after 3 months the prostheses was constructed by using digital workflow
  Interventions: Procedure: implant placement
- PFM fixed hybrid prostheses (Other): 5 implants were placed in mandibular arch by surgical guide and after 3 months the prostheses was constructed by using digital workflow until making wax pattern the casting was made.
  Interventions: Procedure: implant placement

INTERVENTIONS:
Procedure: implant placement — 5 implant were placed in intraforaminal area using surgical guide
  Other Names: final prostheses was made on 5 implants

SUMMARY:
the purposse of the study To evaluate the effect of implant supported hybrid prostheses on the bone of the supporting structure of edentulous mandible using Polyetherketoneketone (PEKK) framework versus cobalt chromium framework. fourteen female patients with lower single edentulous ridges are chosen with adequate dental hygiene, enough interarch space and free of systemic diseases and parafunctional habits. Patients who received new single dentures are randomly allocated into each group using computer software program and five intraforaminal implants were inserted parallel using surgical guide.

DETAILED DESCRIPTION:
Patient's approval:

* All patients will be informed in details about the nature of the investigation and the aim of the study. They will agree to take part in the study and will sign on an informed consent form.
* All participants will be given notice about their privacy practices, their legal duties and their rights.
* In case of implant treatment failure, the patients will receive a new well-fitting denture.

Patient's grouping:

In this study there will be two equal groups, grouping will be based on the material that will be used for framework construction:

Group I: framework will be fabricated using PEKK. Group II: frame work will be fabricated using cobalt chromium alloy.

Clinical steps:

Pre-prosthetic phase:-

* Conventional single lower denture will be made for all patients.
* Occlusal adjustment of upper teeth will be done for all patients.
* The single lower denture will be duplicated with radiographic markers and CBCT will be used to determine exact position of implants.

Surgical phase:-

* Five conventional implants in intraforaminal area will be placed according to the planned cone beam CT using surgical guide to accurately place the implants.
* Postoperative analgesics and anti-inflammatory medications will be described.
* After osseointegration, second surgery will be carried out and healing abutment will be screwed for each implant.

Prosthetic phase:-

* After healing period open top tray impression will be made.
* Jaw relation record will be taken using record bases and wax rims.
* Group I: The PEKK framework will be milled using milling machine.
* Group II: cobalt chromium framework will be made with wax pattern milling then casted by conventional method.
* The PEKK framework will be veneered with zirconia and the cobalt chromium will be veneered with porcelain.
* Implant supported fixed detachable prostheses using PEKK framework or cobalt-chromium framework will be screw retained to conventional implants.

ELIGIBILITY:
Inclusion Criteria:

* Patient's age range from 50 to 60 year's old.
* All patients are with completely edentulous mandible.
* Good oral hygiene is mandatory.
* Sufficient interarch space to accept implant supported fixed prosthesis will be diagnosed by mounted diagnostic casts.
* Firm and healthy mucosa covering the alveolar ridge.
* Minimum bone width 5.5mm buccolinguallly and 10 mm height will be diagnosed by the preoperative cone beam CT scan.

Exclusion Criteria:

* - Vulnerable group; prisoners, mentally, physically disabled, pregnant females.
* Patients with Para functional habits.
* Patients having TMJ disorders.
* Uncontrolled diabetic patients
* Patients have any medical condition or any disease that could interfere with implant placement or affect bone loss.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2023-09-02 (Actual)

PRIMARY OUTCOMES:
amount of bone loss around implant | 2 years
  The points of first bone contact with the fixture platform were detected and changes of those points position through the two years of observation were registered as a criterion of bone changes with further calculation of average values. A software ruler of CBCT was used to measure the crestal bone height in contact with the implant from the four aspects (buccal, lingual, mesial and distal).

CONTACTS AND LOCATIONS:
Overall Officials: dina essam bahig, Principal Investigator — Ain Shams University
Locations (1):
- Dalia Mohammed Farid, Cairo, Egypt